CLINICAL TRIAL: NCT04233411
Title: The Bioavailability of Mycoprotein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 157758
Record Dates: First submitted 2016-11-30; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Availability of Mycoprotein

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Milk (Active Comparator): Acute ingestion of 20 g milk protein
  Interventions: Other: Mycoprotein ingestion
- 20g (Experimental): Acute ingestion of 20 g mycoprotein
  Interventions: Other: Mycoprotein ingestion
- 40g (Experimental): Acute ingestion of 40 g mycoprotein
  Interventions: Other: Mycoprotein ingestion
- 60g (Experimental): Acute ingestion of 60 g mycoprotein
  Interventions: Other: Mycoprotein ingestion
- 80g (Experimental): Acute ingestion of 60 g mycoprotein
  Interventions: Other: Mycoprotein ingestion

INTERVENTIONS:
Other: Mycoprotein ingestion

SUMMARY:
To evaluate the bioavailability of mycoprotein, compared with a reference animal based protein, in a dose-response manner.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and aged 18-40 y
* BMI between 18 and 30

Exclusion Criteria:

* On medication
* Family history of metabolic disease
* Diagnosed with any metabolic or cardiovascular conditions
* BMI < 18 or > 30

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01; Primary Completion 2017-08 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Plasma total amino acid concentrations | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin T Wall, PhD, Principal Investigator — University of Exeter, College of Life and Environmental Sciences
Locations (1):
- Sport & Health Sciences, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No